CLINICAL TRIAL: NCT00069225
Title: Cerebral Structure and Function Before and After Pharmacological and Psychological Treatment for PTSD
Brief Title: Brain Structure and Function Before and After Treatment for Post-Traumatic Stress Disorder
Status: Completed | Type: Observational
Sponsor: National Institute of Mental Health (NIMH) (NIH)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 030297; 03-M-0297
Record Dates: First submitted 2003-09-17; First posted 2003-09-18 (Estimated); Last update posted 2008-03-04 (Estimated); Status verified 2005-09

CONDITIONS: Stress Disorders, Post-Traumatic
Keywords: fMRI; Prolonged Exposure; Brain Activation; Conditioning; Paroxetine; PTSD; Differential Fear Conditioning; Masked Faces; Amygdala; Hippocampus; Post-Traumatic Stress Disorder
MeSH Terms: conditions — Stress Disorders, Post-Traumatic

SUMMARY:
This study, conducted at the University of Pennsylvania and at the National Institutes of Health in Bethesda, Maryland, will examine deficits in brain structure and function in people exposed to trauma who developed post-traumatic stress disorder (PTSD) to see if these deficits change after treatment. It also will investigate whether there is a genetic susceptibility to PTSD.

Candidates 18 years of age and older in the following categories will be included in this study: 1) women who have PTSD of at least 1 year's duration following sexual or non-sexual assault; 2) healthy women (controls) who were previously assaulted but did not develop PTSD; and 3) healthy women (controls) who were never traumatized. Candidates will be screened with a medical history and physical examination, psychiatric evaluation, electrocardiogram (EKG), and routine blood and urine tests.

Women with PTSD will be assigned to receive either: 1) 12 weeks of cognitive behavioral psychotherapy either immediately upon enrollment or after a 3-month waiting period; or 2) 10 weeks of drug treatment with paroxetine (Paxil® (Registered Trademark)). Patients will be evaluated before and after treatment with the procedures outlined below. Control subjects will undergo the same procedures, also with a 10- to 12-week interval between evaluations.

* Neuropsychological testing: Subjects will take paper and pencil and computer tests to evaluate memory, learning, attention and concentration, vocabulary and naming.
* Magnetic resonance imaging (MRI): Subjects will have MRI scans of the brain to examine brain structure and blood flow while they perform two tasks. In the first task, they will be shown a series of faces and asked to press one button for a male face and another button for a female face. In the second task they will hear loud noises and see colored squares. During the scan, subjects lie on a bed that slides into a narrow tunnel (the scanner). They will wear a headset to block the noise of the scanner and through which they will receive instructions for the tasks. Heart rate and skin conductance (sweating) will be measured during the scan to evaluate physiologic changes in response to the tasks.
* Eyeblink air puff test: Subjects will hear tones and will have a light puff of air delivered to the eye. Changes in heart rate, sweat, and eyeblink will be measured with electrodes taped to the skin on two fingers, on each side of the rib cage, and under one eye.
* Potential air puff delivery: This experiment has three parts. During each of the three parts of this experiment, subjects will see colored lights and may or may not receive a puff of air to the neck. Before each part they will be told that they will, will not, or may receive an air puff to the neck. Each part will be repeated several times. During the test, electrodes will be taped to the arms and chest to monitor skin conductance and heart rate responses.
* Blood draw for genetic evaluation: Subjects' DNA will be examined to try to determine if the risk of developing PTSD is inherited. The DNA will be examined for cortisol receptor gene evaluation, to see if a form of this gene is found more often in patients with PTSD than in healthy controls. The receptor for cortisol determines the activity of the stress hormone cortisol, and genetic variations in the structure of this receptor may be related to vulnerability to PTSD.

Patients taking paroxetine will be offered up to 3 months of additional drug therapy following completion of the study and will be offered participation in other NIH studies for evaluation and treatment of PTSD.

DETAILED DESCRIPTION:
Posttraumatic stress disorder (PTSD) is characterized by intrusive recollections, avoidant behavior, anxiety and exaggerated fear response. The pathophysiology of PTSD is largely unknown. Neurophysiological testing in PTSD reveals deficits in memory and attention. Neuroimaging studies report increased amygdala and decreased anterior cingulate activation and reduced hippocampal volume. Clinical observations, psychophysiological measures and animal studies suggest that facilitated fear conditioning, delayed extinction, inescapable shock, sensitization and protracted habituation may contribute to the onset and persistence of PTSD.

We propose to use fMRI and the psychophysiology lab to examine the effect of treatment with paroxetine and cognitive behavioral therapy on regional cerebral blood flow (rCBF) in brain regions conceivably involved in evolution and maintenance of PTSD: Amygdala, anterior cingulate and hippocampus. We will use emotional tasks that have elicited differences in perfusion or metabolism between patients with PTSD and trauma exposed and healthy subjects. Tasks performed in the fMRI will include 'masked' and 'unmasked' emotional faces paradigms and differential delay conditioning. Contextual fear provocation and eyeblink trace conditioning will be done in the psychophysiology lab. This evaluation will be performed before and after a 10-week period of treatment with paroxetine and a 10-session course of cognitive behavioral treatment (CBT).

Study population will comprise the following matched groups: Patients with PTSD; previously traumatized healthy subjects who have not suffered from PTSD and non-traumatized healthy subjects. Subjects from the 1st group will either be treated with paroxetine for 10 weeks, undergo a 10-week 'prolonged exposure' (PE) CBT course, or will be put on the 'waiting list'. It is assumed that variability in outcome will be observed in both treatment modes, which will enable us to seek treatment response predictors.

It is unknown whether cerebral abnormalities in PTSD are state or trait phenomena. In depression and OCD, functional imaging research shows improvement in malfunctioning brain regions after clinically effective psychopharmacological and psychotherapeutic interventions and after administration of placebo in depression. An increase in hippocampal volume was found in patients with PTSD after treatment with paroxetine and after correction of the endocrine abnormality in Cushing's disorder. These findings support our expectation that at least some brain abnormalities in PTSD are state related, and that change in these abnormalities is demonstrable by fMRI.

ELIGIBILITY:
INCLUSION CRITERIA:

Men and women aged 18-65, suffering from PTSD, healthy trauma survivors and never traumatized healthy subjects. PTSD diagnosis will be determined using the structured clinical interview for DSM IV (SCID)(155).

Capable of providing informed consent, obtained prior to any study procedures.

Free of all psychotropic medication for at least 2 weeks, excluding short-term hypnotics. Patients who were treated with fluoxetine will only be included after a medication free period of at least 8 weeks.

Good physical health, confirmed by a complete physical exam (including normal vital signs), electrocardiogram, neurological exam, and routine laboratory tests of blood and urine. However, if patients have participated in other research studies or have had blood work through their primary MD within the last 6 months, these results will be used instead of repeating blood draws for inclusion into the study.

Right handed, as determined by a handedness questionnaire.

EXCLUSION CRITERIA:

Past head trauma involving loss of consciousness, or amnesia greater than 24 hours. This magnitude of head trauma could contribute to psychopathology and brain structure in a manner different than PTSD thereby confounding results.

Substance abuse (alcohol or drugs) or dependence within 3 months prior to screening. The effect of abuse/dependence on phenomenology and biology could mask and exceed PTSD effect.

All additional DSM IV Axis I comorbidity, excluding secondary diagnoses of major depressive disorder (MDD) or anxiety disorders (AD). Given the high comorbidity of these disorders in PTSD, and since excluding such patients would not provide the full spectrum of the disorder, only patients in whom axis I diagnoses of MDD and AD preceded onset of PTSD will be excluded.

Mental retardation or another pervasive developmental disorder.

Risk of homicide or suicide.

When the trauma involves assault, a continuing intimate relationship with the perpetrator.

Current or intended pregnancy. If a participant becomes pregnant during the course of the study, her data will be removed from the analyses.

Subjects who are doing well on medication. Although we will only recruit non-medicated patients, the decision to stop medication will be taken purely on clinical grounds. No subject will be taken off medication solely to participate in the study.

Deafness will NOT exclude patients or healthy controls from participation. Accomodations and protocol adjustments (e.g., abbreviation of neuropsychological battery to eliminate tests which would be subjected to known or expected normalization violations) will be made as necessary for this population.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 95
Dates: Start 2003-09; Study Completion 2005-09

CONTACTS AND LOCATIONS:
Locations (1):
- National Institute of Mental Health (NIMH), Bethesda, Maryland, United States

REFERENCES:
- [Background] Martin SD, Martin E, Rai SS, Richardson MA, Royall R. Brain blood flow changes in depressed patients treated with interpersonal psychotherapy or venlafaxine hydrochloride: preliminary findings. Arch Gen Psychiatry. 2001 Jul;58(7):641-8. doi: 10.1001/archpsyc.58.7.641. PMID 11448369
- [Background] Brody AL, Saxena S, Stoessel P, Gillies LA, Fairbanks LA, Alborzian S, Phelps ME, Huang SC, Wu HM, Ho ML, Ho MK, Au SC, Maidment K, Baxter LR Jr. Regional brain metabolic changes in patients with major depression treated with either paroxetine or interpersonal therapy: preliminary findings. Arch Gen Psychiatry. 2001 Jul;58(7):631-40. doi: 10.1001/archpsyc.58.7.631. PMID 11448368
- [Background] Baxter LR Jr, Schwartz JM, Bergman KS, Szuba MP, Guze BH, Mazziotta JC, Alazraki A, Selin CE, Ferng HK, Munford P, et al. Caudate glucose metabolic rate changes with both drug and behavior therapy for obsessive-compulsive disorder. Arch Gen Psychiatry. 1992 Sep;49(9):681-9. doi: 10.1001/archpsyc.1992.01820090009002. PMID 1514872